CLINICAL TRIAL: NCT07302061
Title: "Effects of Fluid Status and Regional Cerebral Oxygenation on Postoperative Cognitive Dysfunction in Patients Undergoing Lower Extremity Surgery Under General and Spinal Anesthesia."
Acronym: AECGSKD002
Status: Active, not recruiting | Type: Observational
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aygul Valiyeva, research assistant, Goztepe Training and Research Hospital
Other Study IDs: AECGSKD002
Record Dates: First submitted 2025-08-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Cognitive Deficit (POCD)
Keywords: POCD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- General Anesthesia
- Spinal anesthesia

SUMMARY:
We frequently encounter cognitive impairments in patients over 65 undergoing Lower extremity surgery, depending on comorbidities and the choice of anesthesia method. The current development of neuraxial anesthesia techniques and close monitoring devices helps us prevent and detect cognitive impairment early in these patients. In this study, we aimed to investigate the effects of different anesthesia techniques (general anesthesia/spinal anesthesia) applied in orthopedic cases on patient fluid status (pleth variablity index) and regional cerebral oxygenation (NIRS), and their relationship with cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 65
* Patients with an American Society of Anesthesiologists (ASA) score of II-III
* Patients with a Mini Mental State Examination (MMSE) score of ≥24 on the first day before surgery

Exclusion Criteria:

* Patients with coagulation disorders
* Patients with a history of anticoagulant medication use
* Patients with advanced organ failure
* Patients with Alzheimer's disease or advanced dementia
* Patients with allergies to the medications used in the study
* Mental Retardation
* Patients with a wound infection at the site of spinal anesthesia
* Patients with a history of cerebrovascular hemorrhage
* Patients who did not consent;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing Lower extremity surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Early postoperative period (24th and 48th hours) cognitive dysfunction rate | Up to 48 hours after operation
  We will assess postoperative cognitive dysfunction.Cognitive function will be evaluated using the MOCA (Montreal Cognitive Assessment) at 24 and 48 hours after surgery.

SECONDARY OUTCOMES:
Pleth Variability Index (PVI, %) to assess intraoperative fluid status | During Surgery
  PVI values will be continuously recorded using non-invasive monitor.

OTHER OUTCOMES:
Mini Mental State Examination (MMSE) | Up to 48 hours
  Mini Mental State Examination (MMSE) will be recorded as the secondary supportive measure like MOCA.

CONTACTS AND LOCATIONS:
Locations (1):
- Goztepe training and research hospital, Istanbul, Kadikoy, Turkey (Türkiye)